CLINICAL TRIAL: NCT03064347
Title: Targeted Enteral Nutrient Delivery: A Prospective Randomized Study
Acronym: TEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Beale, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TEND HS-16-00339
Record Dates: First submitted 2017-02-17; First posted 2017-02-27 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Obesity; Nutrient
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Sucrose; Whey Proteins; Pea Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Coated Sucrose plus Whole Milk (Active Comparator): 200kcal sucrose plus whole milk powder in enteric coating as single dose
  Interventions: Dietary Supplement: Sucrose plus Whole Milk Powder in Enteric Coating
- Non Coated Sucrose plus Whole Milk (Placebo Comparator): 200kcal sucrose plus whole milk powder with separate enteric coating materials as single dose
  Interventions: Dietary Supplement: Non coated Sucrose plus Whole Milk
- Enteric Coated Sucrose (Active Comparator): 200kcal sucrose in enteric coating as single dose
  Interventions: Dietary Supplement: Sucrose in Enteric Coating
- Non-Enteric Coated Sucrose (Placebo Comparator): 200kcal sucrose with separate enteric coating materials as single dose
  Interventions: Dietary Supplement: Sucrose with Separate Enteric Coating Materials
- Enteric Coated Whey Protein (Active Comparator): 200kcal whey protein in enteric coating as single dose
  Interventions: Dietary Supplement: Whey Protein in Enteric Coating
- Non-Enteric Coated Whey Protein (Placebo Comparator): 200kcal whey protein with separate enteric coating materials as single dose
  Interventions: Dietary Supplement: Whey Protein with Separate Enteric Coating Materials
- Enteric Coated Pea Protein (Active Comparator): 200kcal pea protein in enteric coating as single dose
  Interventions: Dietary Supplement: Pea Protein in Enteric Coating
- Non-Enteric Coated Pea Protein (Placebo Comparator): 200kcal pea protein with separate enteric coating materials as single dose
  Interventions: Dietary Supplement: Pea Protein with Separate Enteric Coating Materials

INTERVENTIONS:
Dietary Supplement: Sucrose plus Whole Milk Powder in Enteric Coating — Single dose enteric coated sucrose plus whole milk powder will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Coated Sucrose plus Whole Milk
Dietary Supplement: Non coated Sucrose plus Whole Milk — Single dose sucrose plus whole milk powder with separate enteric coating materials will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Non Coated Sucrose plus Whole Milk
Dietary Supplement: Sucrose in Enteric Coating — Single dose enteric coated sucrose will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Enteric Coated Sucrose
Dietary Supplement: Sucrose with Separate Enteric Coating Materials — Single dose sucrose with separate enteric coating materials will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Non-Enteric Coated Sucrose
Dietary Supplement: Whey Protein in Enteric Coating — Single dose enteric coated whey protein will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Enteric Coated Whey Protein
Dietary Supplement: Whey Protein with Separate Enteric Coating Materials — Single dose whey protein with separate enteric coating materials will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Non-Enteric Coated Whey Protein
Dietary Supplement: Pea Protein in Enteric Coating — Single dose enteric coated pea protein will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Enteric Coated Pea Protein
Dietary Supplement: Pea Protein with Separate Enteric Coating Materials — Single dose pea protein with separate enteric coating materials will be consumed by mouth. Blood will be drawn at baseline and then at 15 minute intervals for 3 hours from ingestion for measurement of GLP-1, PYY, C-peptide, insulin and glucose.Visual analog score will be used to record satiety and adverse symptoms every 15 minutes.
  Arms: Non-Enteric Coated Pea Protein

SUMMARY:
This study will evaluate whether enteric-coated nutrients increase some glucose and regulating hormone levels, glucose tolerance and satiety in overweight and obese individuals with type 2 diabetes.

DETAILED DESCRIPTION:
Direct delivery of nutrient to the upper intestine by enteral feeding tube can increase circulating levels of some glucose and appetite regulating hormones when compared to usual oral ingestion. Such an enhancement could be of value in the management of type 2 diabetes and obesity. In this study enteric-coated nutrients will be ingested to allow for direct delivery of nutrient to the upper intestine. Levels of select hormones and glucose, and measures of satiety and adverse effects will be compared following the ingestion of uncoated and enteric coated nutrient.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* BMI >27kg/m2
* Type 2 diabetes with known duration of <10years
* On metformin, sulfonylureas, thiazolidinedione or SGLT2 inhibitor or lifestyle management alone or in combination only for management of type 2 diabetes

Exclusion Criteria:

Conditions

* Known foregut pathology or prior foregut surgery.
* Previous surgical treatment for obesity (excluding liposuction if performed > one year before trial entry)
* Known cardiovascular disease other than controlled hypertension
* Known proliferative retinopathy or maculopathy requiring acute treatment, as judged by the Investigator
* Known untreated or uncontrolled hypothyroidism/hyperthyroidism
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Obesity induced by other endocrinologic disorders (e.g. Cushing Syndrome)
* Cancer (past or present except basal cell skin cancer or squamous cell skin cancer), which in the Investigator's opinion could interfere with the results of the trial
* Use of insulin, DPP4 inhibitors or GLP-1 analogs in the previous 1 month
* Treatment with any antidiabetic agent(s) other than metformin, sulphonylurea thiazolidinedione or SGLT-2 inhibitors in the 1 month prior to screening
* Use of any drug (except for metformin, sulphonylurea or thiazolidinedione or SGLT-2 inhibitors), which in the Investigator's opinion could interfere with glucose level (e.g. systemic corticosteroids)
* Receipt of any other anti-diabetic investigational drug within 1 month prior to screening for this trial, or receipt of any investigational drugs not affecting diabetes within 1 month prior to screening for this trial
* Current or history of treatment with medications that may cause significant weight gain, within 1 month prior to screening for this trial, including systemic corticosteroids (except for a short course of treatment, i.e., 7- 10 days), tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g., imipramine, amitryptiline, mirtazapin, paroxetine, phenelzine, clorpromazine, olanzapine,valproic acid and its derivatives, and lithium) thioridazine, clozapine,
* Currently using or have used within three months prior to screening for this trial: pramlintide, sibutramine, orlistat, zonisamide, topiramate or phenteremine (either by prescription or as part of a clinical trial)
* Simultaneous participation in any other clinical trial of an investigational drug
* The receipt of any investigational product within four weeks prior to screening for this trial Herbal supplements or over-the-counter medications
* Diet attempts using herbal supplements or over-the-counter medications within 1 month prior to screening into this trial Other
* Milk allergy
* Lactose intolerance Language barrier, mental incapacity, unwillingness or inability to understand and be able to complete the study Females of childbearing potential
* Pregnant breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by US: abstinence and the following methods: diaphragm with spermacide, condom with spermacide (by male partner), intrauterine device, sponge, spermacide, Norplant®, Depo-Provera® or oral contraceptives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Difference in AUC of GLP-1 on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of blood GLP-1 on meal tolerance tests.

SECONDARY OUTCOMES:
Difference in Peak PYY on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of blood PYY on 3 hour meal tolerance test
Difference in Peak C-peptide on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of blood C-peptide on 3 hour meal tolerance test
Difference in Peak insulin on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of blood insulin on 3 hour meal tolerance test
Difference in Peak glucose on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of blood glucose on 3 hour meal tolerance test
Difference in Peak satiety on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of satiety on 3 hour meal tolerance test measured on a 15mm visual analog scale
Difference in Peak Adverse Events on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of adverse symptoms on 3 hour meal tolerance test measured on a 15mm visual analog scale
Difference in AUC of PYY on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of blood PYY on meal tolerance tests.
Difference in AUC of C-peptide on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of blood C-peptide on meal tolerance tests.
Difference in AUC of insulin on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of blood insulin on meal tolerance tests.
Difference in AUC of glucose on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of blood glucose on meal tolerance tests.
Difference in AUC of satiety on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of satiety on meal tolerance tests of adverse symptoms on 3 hour meal tolerance test measured on a 15mm visual analog scale
Difference in AUC of adverse symptoms on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Integrated Area under the curve (AUC) levels of adverse symptoms on meal tolerance tests of adverse symptoms on 3 hour meal tolerance test measured on a 15mm visual analog scale
Difference in Peak GLP-1 on meal tolerance tests Enteric Coated vs. Uncoated Nutrient. | From ingestion to 3 hours post ingestion.
  Highest level of blood GLP-1 on 3 hour meal tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Beale, MD, Principal Investigator — University of Southern California, Keck School of Medicine
Locations (1):
- USC Diabetes & Obesity Research Institute (DORI), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No